CLINICAL TRIAL: NCT03684694
Title: A Phase 1/2 Open-Label Study to Evaluate the Safety and Efficacy of Loncastuximab Tesirine and Ibrutinib in Patients With Advanced Diffuse Large B-Cell Lymphoma or Mantle Cell Lymphoma (LOTIS-3)
Brief Title: Safety and Efficacy Study of Loncastuximab Tesirine + Ibrutinib in Diffuse Large B-Cell or Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Administrative decision
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-103; 2018-002625-38 (EudraCT Number)
Record Dates: First submitted 2018-09-11; First posted 2018-09-26 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma
Keywords: Loncastuximab Tesirine in Combination with Ibrutinib
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — loncastuximab tesirine; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Dose-Escalation of ADCT-402 (Experimental): A standard 3+3 dose escalation design will be used. The dose-limiting toxicity (DLT) period will be the 21 days following the first dose of ibrutinib. The dose escalation cohort will receive loncastuximab tesirine for Cycle 1 and 2 (3 weeks each) with concurrent ibrutinib (concomitant therapy) daily. Participants may continue to receive ibrutinib therapy up to 1 year after Cycle 1 Day 1 (once every 4 weeks from Cycle 3 onwards). Loncastuximab tesirine will be administered intravenously (IV).
  Interventions: Drug: Loncastuximab Tesirine; Drug: Ibrutinib
- Phase 2: MTD or RP2D of ADCT-402 in Non-GCB DLBCL (Experimental): Participants with non-germinal center B-cell diffuse large B-cell lymphoma (Non-GCB DLBCL) will receive the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of loncastuximab tesirine, as determined in Phase 1, once every 3 weeks for Cycle 1 and 2 and a daily dose of ibrutinib. Participants can continue treatment up to 1 year (once every 4 weeks from Cycle 3 onwards). Loncastuximab tesirine will be administered IV.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Ibrutinib
- Phase 2: MTD or RP2D of ADCT-402 in GCB DLBCL (Experimental): Participants with germinal center B-cell diffuse large B-cell lymphoma (GCB DLBCL) will receive the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of loncastuximab tesirine, as determined in Phase 1, once every 3 weeks for Cycle 1 and 2 and a daily dose of ibrutinib. Participants can continue treatment up to 1 year (once every 4 weeks from Cycle 3 onwards). Loncastuximab tesirine will be administered IV.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Ibrutinib
- Phase 2: MTD or RP2D of ADCT-402 in MCL (Experimental): Participants with mantle cell lymphoma (MCL) will receive the maximum tolerated dose (MTD) or recommended Phase 2 dose (RP2D) of loncastuximab tesirine, as determined in Phase 1, once every 3 weeks for Cycle 1 and 2 and a daily dose of ibrutinib. Participants can continue treatment up to 1 year (once every 4 weeks from Cycle 3 onwards). Loncastuximab tesirine will be administered IV.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Ibrutinib

INTERVENTIONS:
Drug: Loncastuximab Tesirine — Intravenous (IV) infusion.
  Other Names: Zynlonta; ADCT-402
Drug: Ibrutinib — Oral capsule.

SUMMARY:
The purpose of this Phase 1/2 study is to evaluate the safety and efficacy of Loncastuximab Tesirine (ADCT-402) in combination with Ibrutinib in participants with Advanced Diffuse Large B-Cell Lymphoma or Mantle Cell Lymphoma.

DETAILED DESCRIPTION:
The Phase 1 portion of the study will cover the dose escalation portion of the study. This will then be followed by the Phase 2 portion of the study, which will treat participants with the dose of loncastuximab tesirine determined in the Phase 1 portion of the study. The ibrutinib dose of 560 mg daily, will remain the same throughout both phases of the study.

A standard 3+3 dose escalation design will be used for the Phase 1 portion of the study. The dose-limiting toxicity (DLT) period will be the 21 days following the first dose of ibrutinib. The dose escalation cohort will receive loncastuximab tesirine for 2 cycles with concurrent ibrutinib (concomitant therapy) and may then continue ibrutinib therapy up to one year.

The Phase 2 portion of the study will involve 3 cohorts:

* Non-germinal center B-cell diffuse large B-cell lymphoma (Non-GCB DLBCL) cohort
* Germinal center B-cell diffuse large B-cell lymphoma (GCB DLBCL) cohort
* Mantle cell lymphoma (MCL) cohort

Each of the cohorts will be treated with the recommended dose of loncastuximab tesirine determined in the Phase 1 portion of the study.

The study will include a Screening Period (of up to 28 days), a Treatment Period (cycles of 3 to 4 weeks), and a Follow-up Period (approximately every 12 week visits for up to 2 years after treatment discontinuation).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant aged 18 years or older
2. Pathologic diagnosis of DLBCL or MCL (For Italy Sites Only: MCL patients are excluded.)
3. Participants with DLBCL must have relapsed or refractory disease and have failed or been intolerant to available standard therapy
4. Participants with MCL must have relapsed or refractory disease and have received at least one prior line of therapy (For Italy Sites Only: This exclusion criterion is not applicable)
5. Participants who have received previous CD19-directed therapy must have a biopsy which shows CD19 expression after completion of the CD19-directed therapy
6. Measurable disease as defined by the 2014 Lugano Classification
7. Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block (or minimum 10 freshly cut unstained slides if block is not available)
8. ECOG performance status 0 to 2
9. Screening laboratory values within the following parameters:

   1. Absolute neutrophil count (ANC) ≥1.0 × 103/µL (off growth factors at least 72 hours)
   2. Platelet count ≥75 × 103/µL without transfusion in the past 7 days
   3. Hemoglobin ≥8 g/dL (4.96 mmol/L), transfusion allowed
   4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and gamma glutamyl transferase (GGT) ≤2.5 × the ULN
   5. Total bilirubin ≤1.5 × ULN (participants with known Gilbert's syndrome may have a total bilirubin up to ≤3 × ULN)
   6. Blood creatinine ≤1.5 × ULN or calculated creatinine clearance ≥60 mL/min by the Cockcroft and Gault equation
10. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test within 7 days prior to start of study drugs on C1D1 for women of childbearing potential
11. Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 9 months after the last dose of loncastuximab tesirine or 1 month after last dose of ibrutinib, whichever comes last. Men with female partners who are of childbearing potential must agree that they will use a highly effective method of contraception from the time of giving informed consent until at least 6 months after the participant receives his last dose of loncastuximab tesirine or 3 months after last dose of ibrutinib, whichever comes last

Exclusion Criteria:

1. Known history of hypersensitivity to or positive serum human anti-drug antibody (ADA) to a CD19 antibody
2. Known history of hypersensitivity to ibrutinib
3. Previous therapy with ibrutinib or other BTK inhibitors
4. Previous therapy with loncastuximab tesirine
5. Requires treatment or prophylaxis with a moderate or strong cytochrome P450 (CYP) 3A inhibitor
6. Allogenic or autologous transplant within 60 days prior to start of study drugs (C1D1)
7. Active graft-versus-host disease
8. Post-transplantation lymphoproliferative disorder
9. Active autoimmune disease, including motor neuropathy considered of autoimmune origin and other central nervous system (CNS) autoimmune disease
10. Known seropositive and requiring anti-viral therapy for human immunodeficiency (HIV) virus, hepatitis B virus (HBV), or hepatitis C virus (HCV).
11. History of Stevens-Johnson syndrome or toxic epidermal necrolysis
12. Lymphoma with active CNS involvement at the time of screening, including leptomeningeal disease
13. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
14. Breastfeeding or pregnant
15. Significant medical comorbidities, including but not limited to, uncontrolled hypertension (blood pressure [BP] ≥160/100 millimeters of mercury (mmHg) repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 6 months prior to screening, uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes mellitus, or severe chronic pulmonary disease, or tuberculosis infection (tuberculosis screening based on local standards).
16. Major surgery, radiotherapy, chemotherapy, or other anti-neoplastic therapy within 14 days prior to start of study drugs (C1D1), except shorter if approved by the Sponsor
17. Use of any other experimental medication within 14 days prior to start of study drugs (C1D1)
18. Planned live vaccine administration after starting study drugs (C1D1)
19. Any condition that could interfere with the absorption or metabolism of ibrutinib including malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel
20. Inherited or acquired bleeding disorders
21. Ongoing anticoagulation treatment, except for low-dose heparinisation or equivalent
22. Failure to recover to Grade ≤1 (Common Terminology Criteria for Adverse Events [CTCAE] version 4.0) from acute non-hematologic toxicity (Grade ≤2 neuropathy or alopecia) due to previous therapy prior to screening
23. Congenital long QT syndrome or a corrected QTcF interval of >480 ms at screening (unless secondary to pacemaker or bundle branch block)
24. Active second primary malignancy other than non-melanoma skin cancers, non metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree, and document should not be exclusionary
25. Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgement, make the participant inappropriate for study participation or put the participant at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (12):
  - University of California Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - Redlands Community Hospital, Redlands, California
  - University of Miami, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - The Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Vincent Healthcare, Billings, Montana
  - Case Western Reserve University, Cleveland, Ohio
- Belgium (2):
  - GasthuisZusters Antwerpen Sint-Augustinus, Wilrijk
  - CHU UCL Namur (Site Godinne), Yvoir
- France (6):
  - Centre Hospitalier Universitaire de Rennes Hôpital Pontchailou, Bretagne
  - Hôpital Hôtel-Dieu, Loiré
  - Hôpital Saint-Eloi, Montpellier
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire De Poitier - Hopital De La Miletrie - Hopital Jean Bernard, Poitiers
- Italy (7):
  - IRCCS istituto Clinico Humanitas U.O. di Oncologia ed Ematologia, Via Manzoni, Rozzano
  - Azienda Ospedaliera Pap Giovanni XXIII, Bergamo
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Istituto Scientifico Rmagnolo per lo Studio e la Cura dei Tumori, Meldola FC
  - Istituto Europeo di Oncologia, Milan
  - Azienda Unita Sanitaria Locale de Ravenna, Ravenna
- Spain (6):
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Duran I Reynals, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - Abertawe Bro Morgannwg University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 136 participants were enrolled into sites in the United States, Belgium, France, Italy, and Spain.
Pre-assignment Details: Participants were screened for eligibility to enroll within 28 days prior to the start of treatment.
Groups:
- Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib: Participants with advanced diffuse large B-Cell lymphoma (DLBCL) or mantle cell lymphoma (MCL) were enrolled to receive 60 µg/kg of loncastuximab tesirine via intravenous (IV) infusion once every 3 weeks (Q3W) for 2 treatment cycles (cycle is 3 weeks for Cycles 1 and 2) with concurrent 560 mg ibrutinib orally via capsules once daily. Participants who had a response of partial response (PR) or stable disease (SD) at the 14-week assessment may have received 2 additional doses of loncastuximab tesirine given 4 weeks apart on Day 1 of Cycles 5 and 6.
- Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib: Participants with advanced DLBCL or MCL were enrolled to receive 75 µg/kg of loncastuximab tesirine via IV infusion Q3W for 2 treatment cycles (cycle is 3 weeks for Cycles 1 and 2) with concurrent 560 mg ibrutinib orally via capsules once daily. Participants who had a response of PR or SD at the 14-week assessment may have received 2 additional doses of loncastuximab tesirine given 4 weeks apart on Day 1 of Cycles 5 and 6.
- Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib: Participants with advanced DLBCL or MCL were enrolled to receive 90 µg/kg of loncastuximab tesirine via IV infusion Q3W for 2 treatment cycles (cycle is 3 weeks for Cycles 1 and 2) with concurrent 560 mg ibrutinib orally via capsules once daily. Participants who had a response of PR or SD at the 14-week assessment may have received 2 additional doses of loncastuximab tesirine given 4 weeks apart on Day 1 of Cycles 5 and 6.
- Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL: Participants with non-germinal center B-cell (GCB) DLBCL received the recommended phase 2 dose (RP2D) of 60 µg/kg loncastuximab tesirine via IV infusion with concurrent 560 mg ibrutinib orally via capsules once daily. Loncastuximab tesirine was administered on Day 1 of Cycles 1 and 2 (cycle is 3 weeks for Cycles 1 and 2, and 4 weeks for Cycles 3 onwards). Participants who had a response of complete response (CR), PR, and SD received additional doses of loncastuximab tesirine on Day 1 of Cycles 5, 6, 9 and 10.
- Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL: Participants with GCB DLBCL received the RP2D of 60 µg/kg loncastuximab tesirine via IV infusion with concurrent 560 mg ibrutinib orally via capsules once daily. Loncastuximab tesirine was administered on Day 1 of Cycles 1 and 2 (cycle is 3 weeks for Cycles 1 and 2, and 4 weeks for Cycles 3 onwards). Participants who had a response of CR, PR, and SD received additional doses of loncastuximab tesirine on Day 1 of Cycles 5, 6, 9 and 10.
- Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL: Participants with MCL received the RP2D of 60 µg/kg loncastuximab tesirine via IV infusion with concurrent 560 mg ibrutinib orally via capsules once daily. Loncastuximab tesirine was administered on Day 1 of Cycles 1 and 2 (cycle is 3 weeks for Cycles 1 and 2, and 4 weeks for Cycles 3 onwards). Participants who had a response of CR, PR, and SD received additional doses of loncastuximab tesirine on Day 1 of Cycles 5, 6, 9 and 10.
Period: Phase 1
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Started | 37 | 4 | 6 | 0 (Participants were not enrolled into the Phase 1 part.) | 0 (Participants were not enrolled into the Phase 1 part.) | 0 (Participants were not enrolled into the Phase 1 part.)
Completed | 0 | 1 | 1 | 0 (Participants were not enrolled into the Phase 1 part.) | 0 (Participants were not enrolled into the Phase 1 part.) | 0 (Participants were not enrolled into the Phase 1 part.)
Not Completed | 37 | 3 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator/Sponsor Decision | 12 | 2 | 1 | 0 | 0 | 0
Not completed — Death | 24 | 0 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Miscellaneous | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Started | 0 (Participants were not enrolled into the Phase 2 part.) | 0 (Participants were not enrolled into the Phase 2 part.) | 0 (Participants were not enrolled into the Phase 2 part.) | 49 | 30 | 10
Completed | 0 (Participants were not enrolled into the Phase 2 part.) | 0 (Participants were not enrolled into the Phase 2 part.) | 0 (Participants were not enrolled into the Phase 2 part.) | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 49 | 30 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Investigator/Sponsor Decision | 0 | 0 | 0 | 17 | 16 | 6
Not completed — Death | 0 | 0 | 0 | 28 | 14 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Measured in the safety analysis set, which included all participants who received study drug.
Groups:
- Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib: Participants with advanced DLBCL or MCL were enrolled to receive 75 µg/kg of loncastuximab tesirine via IV infusion Q3W for 2 treatment cycles (cycle is 3 weeks for Cycles 1 and 2) with concurrent 560 mg ibrutinib orally via capsules once daily. Participants who had a response of partial response (PR) or stable disease (SD) at the 14-week assessment may have received 2 additional doses of loncastuximab tesirine given 4 weeks apart on Day 1 of Cycles 5 and 6.
- Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib: Participants with advanced DLBCL or MCL were enrolled to receive 90 µg/kg of loncastuximab tesirine via IV infusion Q3W for 2 treatment cycles (cycle is 3 weeks for Cycles 1 and 2) with concurrent 560 mg ibrutinib orally via capsules once daily. Participants who had a response of partial response (PR) or stable disease (SD) at the 14-week assessment may have received 2 additional doses of loncastuximab tesirine given 4 weeks apart on Day 1 of Cycles 5 and 6.
- Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL: Participants with non-germinal center B-cell (GCB) DLBCL received the recommended phase 2 dose (RP2D) of 60 µg/kg loncastuximab tesirine via IV infusion with concurrent 560 mg ibrutinib orally via capsules once daily. Loncastuximab tesirine was administered on Day 1 of Cycles 1 and 2 (cycle is 3 weeks for Cycles 1 and 2, and 4 weeks for Cycles 3 onwards). Participants who had a response of complete response (CR), partial response (PR), and stable disease (SD) received additional doses of loncastuximab tesirine on Day 1 of Cycles 5, 6, 9 and 10.
- Total: Total of all reporting groups
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL | Total
Number analyzed (Participants) | 37 | 4 | 6 | 49 | 30 | 10 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 1 | 3 | 13 | 10 | 5 | 43
  >=65 years | 26 | 3 | 3 | 36 | 20 | 5 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 2 | 19 | 9 | 3 | 45
  Male | 27 | 2 | 4 | 30 | 21 | 7 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 0 | 2
  Not Hispanic or Latino | 37 | 4 | 6 | 47 | 27 | 9 | 130
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 2
  White | 35 | 4 | 6 | 43 | 26 | 10 | 124
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 4 | 4 | 0 | 9

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) that occurred or worsened in the period extending from the first dose of study drug to 30 days after the last dose of study drug in this study or start of a new anticancer therapy, whichever is earlier. Any clinically significant changes form baseline in safety laboratory values, vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, and 12-lead electrocardiograms (ECGs) which occurred after first dose of study drug were recorded as TEAEs.
Time Frame: Day 1 until 30 days after last dose; max duration of treatment was 686 days for Phase 1 (up to approximately 716 days total)
Population: Measured in the safety population, which included all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 37 | 4 | 6
Participants | 37 | 4 | 6

2. Primary Outcome: Phase 1: Number of Participants With Serious TEAEs
Description: A serious TEAE was defined as any AE which occurred after the first dose of study drug that resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization (hospitalization for elective procedures or for protocol compliance was not considered a serious adverse event), resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or important medical events that did not meet the preceding criteria but based on appropriate medical judgement may have jeopardized the participant or may have required medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: as for outcome 1
Population: Measured in the safety population, which included all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 37 | 4 | 6
Participants | 19 | 0 | 3

3. Primary Outcome: Phase 1: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following events which occur during the DLT Period (first 21 days of ibrutinib treatment), except those that are clearly due to underlying disease or extraneous causes: a hematologic DLT (grade ≥3 anaemia, grade 4/febrile neutropenia, grade ≥3 thrombocytopenia), a non-hematologic DLT (including aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT] >3× upper limit of normal (ULN) and bilirubin >2× ULN), any other non-hematologic toxicities ≥ Grade 3, with exceptions.
Time Frame: 21 days
Population: Measured in the safety population, which included all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 37 | 4 | 6
Participants | 0 | 0 | 2

4. Primary Outcome: Phase 1: Number of Participants With Dose Interruptions
Time Frame: Up to a maximum of 686 days
Population: Measured in the safety population, which included all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 37 | 4 | 6
Participants | 1 | 0 | 0

5. Primary Outcome: Phase 1: Number of Participants With Dose Reductions
Time Frame: Up to a maximum of 686 days
Population: Measured in the safety population, which included all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 37 | 4 | 6
Participants | 0 | 0 | 0

6. Primary Outcome: Phase 2: Complete Response Rate (CRR)
Description: CRR according to the 2014 Lugano classifications determined by Independent Review Committee (IRC). CRR was defined as the percentage of participants with a best overall response (BOR) of complete response (CR).
Time Frame: Up to approximately 38 months
Population: Measured in the efficacy analysis set, which included all participants who received at least 1 dose of study drug, who had valid baseline disease assessment(s), and who had at least one valid post-baseline disease assessment. Participants who did not have a post-baseline assessment due to early clinical progression or death (after receiving study drug) were also included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 48 | 30 | 10
percentage of participants | 27.1 [15.3 to 41.8] | 26.7 [12.3 to 45.9] | 90.0 [55.5 to 99.7]

7. Secondary Outcome: Phase 1: Overall Response Rate (ORR)
Description: ORR according to the 2014 Lugano classification, defined as the percentage of participants with a BOR of CR or partial response (PR).
Time Frame: Up to approximately 38 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 37 | 4 | 6
percentage of participants | 59.5 [42.1 to 75.2] | 50.0 [6.8 to 93.2] | 50.0 [11.8 to 88.2]

8. Secondary Outcome: Phase 1 and Phase 2: Duration of Response (DOR)
Description: DOR was defined as the time from the first documentation of tumor response to disease progression or death.
Time Frame: Up to approximately 36 months
Population: Measured in the efficacy analysis set, which included all participants who received at least 1 dose of study drug, who had valid baseline disease assessment(s), who had at least one valid post-baseline disease assessment who achieved a response. Participants who did not have a post-baseline assessment due to early clinical progression or death (after receiving study drug) were also included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 22 | 2 | 3 | 23 | 14 | 10
months | 7.49 [2.46 to 20.50] | NA [NA to NA] — Data could not be calculated due to insufficient number of participants with events. | 2.50 [1.94 to NA] — Upper confidence interval could not be calculated due to insufficient number of participants with events. | 8.25 [2.30 to NA] — Upper confidence interval could not be calculated due to insufficient number of participants with events. | 7.64 [1.87 to NA] — Upper confidence interval could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Data could not be calculated due to insufficient number of participants with events.

9. Secondary Outcome: Phase 1 and Phase 2: Relapse-Free Survival (RFS)
Description: RFS was defined as the time from the documentation of CR to disease progression or death.
Time Frame: Up to approximately 36 months
Population: Measured in the efficacy analysis set, which included all participants who received at least 1 dose of study drug, who had valid baseline disease assessment(s), and who had at least one valid post-baseline disease assessment who achieved CR. Participants who did not have a post-baseline assessment due to early clinical progression or death (after receiving study drug) were also included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 15 | 1 | 2 | 13 | 8 | 9
months | 7.49 [3.61 to 22.28] | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events. | 1.94 [NA to NA] — Lower and upper confidence interval could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events.

10. Secondary Outcome: Phase 1 and Phase 2: Progression-Free Survival (PFS)
Description: PFS was defined as the time between start of treatment and the first documentation of progression, or death.
Time Frame: Up to approximately 37 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 37 | 4 | 6 | 48 | 30 | 10
months | 3.55 [1.74 to 7.79] | 3.17 [1.22 to NA] — Upper confidence interval could not be calculated due to insufficient number of participants with events. | 2.12 [0.69 to NA] — Upper confidence interval could not be calculated due to insufficient number of participants with events. | 3.20 [1.41 to 4.99] | 3.02 [1.31 to 6.80] | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events.

11. Secondary Outcome: Phase 1 and Phase 2: Overall Survival (OS)
Description: OS was defined as the time between the start of treatment and death from any cause.
Time Frame: Up to approximately 38 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 37 | 4 | 6 | 48 | 30 | 10
months | 14.23 [7.82 to 25.99] | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events. | 8.54 [4.57 to 20.60] | 16.76 [7.16 to NA] — Upper confidence interval could not be calculated due to insufficient number of participants with events. | NA [NA to NA] — Median, lower and upper confidence interval could not be calculated due to insufficient number of participants with events.

12. Secondary Outcome: Phase 1 and Phase 2: Time to Reach Maximum Concentration (Tmax) of Loncastuximab Tesirine (Total Antibody, PBD-Conjugated Antibody and Unconjugated Cytotoxin SG3199)
Description: Blood samples were collected for analysis of PK data of loncastuximab tesirine (total antibody, PBD-conjugated antibody and unconjugated cytotoxin SG3199)
Time Frame: C1D1 pre-dose, EOI, 4h PD, C1D8 168h PD, C1D15 336h PD, C2D1 pre-dose, EOI, 4h PD, C2D8 168h PD, C2D15 336h PD (3 week cycles)
Population: Measured in the PK population, which included all participants who had at least 1 pre-C1D1 and 1 post-dose valid PK assessment. The "number of participants analzyed" represents the number of participants with collected data. Analysis reported per dose of loncastuximab tesirine as pre-specified.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Groups:
- Phase 1 and Phase 2: 60 µg/kg Loncastuximab Tesirine and Ibrutinib: Participants with advanced diffuse large B-Cell lymphoma (DLBCL) or mantle cell lymphoma (MCL) were enrolled to receive 60 µg/kg of loncastuximab tesirine via intravenous (IV) infusion once every 3 weeks (Q3W) for 2 treatment cycles (cycle is 3 weeks for Cycles 1 and 2) with concurrent 560 mg ibrutinib orally via capsules once daily. Participants in Phase 1 who had a response of partial response (PR) or stable disease (SD) at the 14-week assessment may have received 2 additional doses of loncastuximab tesirine given 4 weeks apart on Day 1 of Cycles 5 and 6. Participants in Phase 2 who had a response of complete response (CR), partial response (PR), and stable disease (SD) received additional doses of loncastuximab tesirine on Day 1 of Cycles 5, 6, 9 and 10.
Arm/Group | Phase 1 and Phase 2: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 124 | 4 | 6
days
  Cycle 1: PBD-conjugated Antibody | 0.0410 (122) | 0.0410 (118) | 0.0330 (108)
  Cycle 1: Total Antibody: number analyzed (Participants) | 122 | 4 | 6
  Cycle 1: Total Antibody | 0.0420 (125) | 0.0410 (118) | 0.0250 (21.1)
  Cycle 1: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 1 | 0 | 1
  Cycle 1: Unconjugated cytotoxin SG3199 | 14.9 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data. |  | 6.94 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data.
  Cycle 2: PBD-conjugated Antibody: number analyzed (Participants) | 113 | 4 | 3
  Cycle 2: PBD-conjugated Antibody | 0.0470 (223) | 0.164 (3347) | 0.0280 (37.8)
  Cycle 2: Total Antibody: number analyzed (Participants) | 110 | 4 | 3
  Cycle 2: Total Antibody | 0.0570 (232) | 0.0370 (136) | 0.0280 (37.8)
  Cycle 2: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 2 | 0 | 0
  Cycle 2: Unconjugated cytotoxin SG3199 | 0.0220 (19.9) |  |

13. Secondary Outcome: Phase 1 and Phase 2: Maximum Observed Concentration (Cmax) of Loncastuximab Tesirine (Total Antibody, PBD-Conjugated Antibody and Unconjugated Cytotoxin SG3199)
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1 and Phase 2: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 124 | 4 | 6
ng/mL
  Cycle 1: PBD-conjugated Antibody | 753 (52.7) | 872 (23.8) | 1065 (17.0)
  Cycle 1: Total Antibody: number analyzed (Participants) | 122 | 4 | 6
  Cycle 1: Total Antibody | 1192 (55.1) | 1270 (29.0) | 2073 (23.5)
  Cycle 1: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 1 | 0 | 1
  Cycle 1: Unconjugated cytotoxin SG3199 | 0.0260 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data. |  | 0.0480 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data.
  Cycle 2: PBD-conjugated Antibody: number analyzed (Participants) | 113 | 4 | 3
  Cycle 2: PBD-conjugated Antibody | 815 (67.0) | 628 (63.1) | 1111 (7.48)
  Cycle 2: Total Antibody: number analyzed (Participants) | 110 | 4 | 3
  Cycle 2: Total Antibody | 1328 (65.0) | 944 (68.8) | 1996 (18.2)
  Cycle 2: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 2 | 0 | 0
  Cycle 2: Unconjugated cytotoxin SG3199 | 0.0450 (85.4) |  |

14. Secondary Outcome: Phase 1 and Phase 2: Area Under the Concentration-Time Curve From Time Zero to the Last Quantifiable Concentration (AUClast) of Loncastuximab Tesirine (Total Antibody, PBD-Conjugated Antibody and Unconjugated Cytotoxin SG3199)
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Phase 1 and Phase 2: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 124 | 4 | 6
day*ng/mL
  Cycle 1: PBD-conjugated Antibody | 3711 (237) | 5899 (34.3) | 5772 (50.0)
  Cycle 1: Total Antibody: number analyzed (Participants) | 122 | 4 | 6
  Cycle 1: Total Antibody | 5528 (244) | 8364 (48.6) | 9877 (56.0)
  Cycle 1: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 1 | 0 | 1
  Cycle 1: Unconjugated cytotoxin SG3199 | 0.105 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data. |  | 0.481 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data.
  Cycle 2: PBD-conjugated Antibody: number analyzed (Participants) | 113 | 4 | 3
  Cycle 2: PBD-conjugated Antibody | 3200 (530) | 5681 (52.4) | 8503 (24.2)
  Cycle 2: Total Antibody: number analyzed (Participants) | 110 | 4 | 3
  Cycle 2: Total Antibody | 4798 (565) | 8828 (63.0) | 15785 (30.0)
  Cycle 2: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 2 | 0 | 0
  Cycle 2: Unconjugated cytotoxin SG3199 | 0.00700 (1118314) |  |

15. Secondary Outcome: Phase 1 and Phase 2: Area Under the Concentration-Time Curve From Time Zero to the End of the Dosing Interval (AUCtau) of Loncastuximab Tesirine (Total Antibody, PBD-Conjugated Antibody and Unconjugated Cytotoxin SG3199)
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Phase 1 and Phase 2: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 78 | 1 | 2
day*ng/mL
  Cycle 1: PBD-conjugated Antibody: number analyzed (Participants) | 0 | 0 | 0
  Cycle 1: Total Antibody: number analyzed (Participants) | 0 | 0 | 0
  Cycle 1: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 0 | 0 | 0
  Cycle 2: PBD-conjugated Antibody | 6785 (55.0) | 6800 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data. | 9084 (26.7)
  Cycle 2: Total Antibody: number analyzed (Participants) | 71 | 1 | 2
  Cycle 2: Total Antibody | 11228 (47.6) | 12419 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data. | 18090 (29.6)
  Cycle 2: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Phase 1 and Phase 2: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUCinf) of Loncastuximab Tesirine (Total Antibody, PBD-Conjugated Antibody and Unconjugated Cytotoxin SG3199)
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | Phase 1 and Phase 2: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 45 | 2 | 3
day*ng/mL
  Cycle 1: PBD-conjugated Antibody | 4766 (47.1) | 5197 (7.00) | 5511 (65.6)
  Cycle 1: Total Antibody: number analyzed (Participants) | 37 | 0 | 3
  Cycle 1: Total Antibody | 8153 (35.6) |  | 11397 (48.8)
  Cycle 1: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 0 | 0 | 0
  Cycle 2: PBD-conjugated Antibody: number analyzed (Participants) | 0 | 0 | 0
  Cycle 2: Total Antibody: number analyzed (Participants) | 0 | 0 | 0
  Cycle 2: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Phase 1 and Phase 2: Clearance (CL) of Loncastuximab Tesirine (Total Antibody, PBD-Conjugated Antibody and Unconjugated Cytotoxin SG3199)
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Phase 1 and Phase 2: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 78 | 2 | 3
L/day
  Cycle 1: PBD-conjugated Antibody: number analyzed (Participants) | 45 | 2 | 3
  Cycle 1: PBD-conjugated Antibody | 0.751 (47.2) | 0.848 (5.00) | 1.06 (96.8)
  Cycle 1: Total Antibody: number analyzed (Participants) | 37 | 0 | 3
  Cycle 1: Total Antibody | 0.548 (34.5) |  | 0.639 (85.2)
  Cycle 1: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 0 | 0 | 0
  Cycle 2: PBD-conjugated Antibody: number analyzed (Participants) | 78 | 1 | 2
  Cycle 2: PBD-conjugated Antibody | 0.548 (51.4) | 0.597 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data. | 0.635 (69.0)
  Cycle 2: Total Antibody: number analyzed (Participants) | 71 | 1 | 2
  Cycle 2: Total Antibody | 0.401 (43.6) | 0.395 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data. | 0.385 (72.6)
  Cycle 2: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Phase 1 and Phase 2: Accumulation Index (AI) Loncastuximab Tesirine (Total Antibody, PBD-Conjugated Antibody and Unconjugated Cytotoxin SG3199)
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1 and Phase 2: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib
Number analyzed (Participants) | 65 | 1 | 2
ratio
  Cycle 1: PBD-conjugated Antibody: number analyzed (Participants) | 0 | 0 | 0
  Cycle 1: Total Antibody: number analyzed (Participants) | 0 | 0 | 0
  Cycle 1: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 0 | 0 | 0
  Cycle 2: PBD-conjugated Antibody | 1.43 (24.6) | 1.15 (NA) — Geometric coefficient of variation could not be calculated as there was only 1 participant with evaluable data. | 1.47 (48.4)
  Cycle 2: Total Antibody: number analyzed (Participants) | 46 | 0 | 2
  Cycle 2: Total Antibody | 1.39 (23.3) |  | 1.36 (33.8)
  Cycle 2: Unconjugated cytotoxin SG3199: number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Phase 1 and Phase 2: Number of Participants With Positive Anti-Drug Antibody (ADA) Titers to Loncastuximab Tesirine at Any Time
Description: Detection of ADAs was performed by using a screening assay for identification of antibody positive samples/participants, a confirmation assay, and titer assessment.
Time Frame: Up to a maximum of 711 days
Population: ADA-evaluable participants including all participants tested for ADAs in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 37 | 4 | 6 | 48 | 29 | 10
Participants | 1 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Phase 2: ORR
Description: ORR according to the 2014 Lugano classification, defined as the percentage of participants with a BOR of CR or PR.
Time Frame: Up to approximately 38 months
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 48 | 30 | 10
percentage of participants | 47.9 [33.3 to 62.8] | 46.7 [28.3 to 65.7] | 100 [69.2 to 100]

21. Secondary Outcome: Phase 2: CRR in Non-GCB DLBCL, GCB DLBCL, All DLBCL and MCL Participants
Description: CRR according to the 2014 Lugano classifications determined by the IRC. CRR was defined as the percentage of participants with a BOR of CR in non-GCB DLBCL, GCB DLBCL, all DLBCL, and MCL participants.
Time Frame: Up to approximately 38 months
Population: Measured in the efficacy analysis set, which included all participants who received at least 1 dose of study drug, who had valid baseline disease assessment(s), and who had at least one valid post-baseline disease assessment. Participants who did not have a post-baseline assessment due to early clinical progression or death (after receiving study drug) were also included. As pre-specified, data are presented for non-GCB DLBCL, GCB DLBCL, all DLBCL, and MCL cohorts.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2: Loncastuximab Tesirine and Ibrutinib in All DLBCL Participants: Participants with all DLBCL types received the RP2D of 60 µg/kg loncastuximab tesirine via IV infusion with concurrent 560 mg ibrutinib orally via capsules once daily. Loncastuximab tesirine was administered on Day 1 of Cycles 1 and 2 (cycle is 3 weeks for Cycles 1 and 2, and 4 weeks for Cycles 3 onwards). Participants who had a response of CR, PR, and SD received additional doses of loncastuximab tesirine on Day 1 of Cycles 5, 6, 9 and 10.
Arm/Group | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in All DLBCL Participants
Number analyzed (Participants) | 48 | 30 | 10 | 78
percentage of participants | 27.1 [15.3 to 41.8] | 26.7 [12.3 to 45.9] | 90.0 [55.5 to 99.7] | 26.9 [17.5 to 38.2]

22. Secondary Outcome: Phase 2: Number of Participants With TEAEs
Description: A TEAE was defined as an adverse event (AE) that occurred or worsened in the period extending from the first dose of study drug to 30 days after the last dose of study drug in this study or start of a new anticancer therapy, whichever is earlier. Any clinically significant changes form baseline in safety laboratory values, vital signs, ECOG performance status, and 12-lead ECGs which occurred after first dose of study drug were recorded as TEAEs.
Time Frame: Day 1 until 30 days after last dose; max duration of treatment was 711 days for Phase 2 (up to approximately 741 days total)
Population: Measured in the safety population, which included all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 49 | 30 | 10
Participants | 48 | 30 | 10

23. Secondary Outcome: Phase 2: Number of Participants With Serious TEAEs
Description: as for outcome 2
Time Frame: as for outcome 22
Population: Measured in the safety population, which included all participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
Number analyzed (Participants) | 49 | 30 | 10
Participants | 27 | 5 | 5

ADVERSE EVENTS:
Time Frame: All-cause mortality reporting was from enrollment until approximately 4 years. For serious adverse events and other adverse events, from Day 1 until 30 days after last dose; max duration of treatment was 686 days for Phase 1 (up to approximately 716 days total), 711 days for Phase 2 (up to approximately 741 days total).
Description: Measured in the safety population, which included all participants who received study drug.
Arm/Group | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL
All-Cause Mortality (participants affected / at risk) | 24/37 | 0/4 | 3/6 | 28/49 | 14/30 | 3/10
Serious Adverse Events (participants affected / at risk) | 19/37 | 0/4 | 3/6 | 27/49 | 5/30 | 5/10
Other Adverse Events (participants affected / at risk) | 37/37 | 4/4 | 6/6 | 48/49 | 30/30 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib (N=37) | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib (N=4) | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib (N=6) | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL (N=49) | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL (N=30) | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL (N=10)
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pericardial disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 2 | 0 | 1 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 4 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 2 | 0 | 0 | 2 | 0 | 1
Citrobacter infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 5 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia parainfluenzae viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 60 µg/kg Loncastuximab Tesirine and Ibrutinib (N=37) | Phase 1: 75 µg/kg Loncastuximab Tesirine and Ibrutinib (N=4) | Phase 1: 90 µg/kg Loncastuximab Tesirine and Ibrutinib (N=6) | Phase 2: Loncastuximab Tesirine and Ibrutinib in Non-Germinal Center B-cell (GCB) DLBCL (N=49) | Phase 2: Loncastuximab Tesirine and Ibrutinib in GCB DLBCL (N=30) | Phase 2: Loncastuximab Tesirine and Ibrutinib in MCL (N=10)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 2 | 4 | 22 | 12 | 4
Anaemia (Blood and lymphatic system disorders) | 9 | 2 | 4 | 13 | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 5 | 3 | 1 | 18 | 7 | 4
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 4 | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 4 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 0 | 2 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 9 | 2 | 1 | 9 | 7 | 5
Nausea (Gastrointestinal disorders) | 9 | 1 | 1 | 5 | 4 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 0 | 6 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 1 | 3 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 5 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1 | 3 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 9 | 0 | 2 | 14 | 2 | 3
Oedema peripheral (General disorders) | 6 | 1 | 1 | 12 | 3 | 1
Asthenia (General disorders) | 6 | 1 | 0 | 5 | 2 | 3
Pyrexia (General disorders) | 2 | 0 | 2 | 10 | 1 | 0
Chills (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 2 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 2 | 0 | 0 | 2 | 1 | 0
Sensation of foreign body (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystocholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypogammaglobulinaemia (Immune system disorders) | 2 | 0 | 0 | 1 | 1 | 0
Conjunctivitis (Infections and infestations) | 6 | 0 | 0 | 1 | 1 | 2
Oral candidiasis (Infections and infestations) | 3 | 0 | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 1 | 3 | 2
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 1
Furuncle (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 1 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 3 | 4 | 3 | 1
Gamma-glutamyltransferase increased (Investigations) | 4 | 0 | 2 | 3 | 2 | 2
Lipase increased (Investigations) | 3 | 0 | 1 | 2 | 2 | 1
Weight increased (Investigations) | 4 | 0 | 0 | 3 | 0 | 0
Weight decreased (Investigations) | 3 | 0 | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 2 | 0 | 0 | 4 | 3 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 3 | 1 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 2 | 0 | 0
Blood iron decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 2 | 5 | 3 | 0
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 1 | 1 | 6 | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0 | 1 | 4 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 0 | 0 | 6 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 7 | 6 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 0 | 0 | 5 | 4 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 2 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 6 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 6 | 0 | 0
Musculoskeletal pain (Metabolism and nutrition disorders) | 2 | 0 | 0 | 4 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 4 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 2 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 0 | 0 | 2 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 4 | 1 | 1
Agitation (Psychiatric disorders) | 2 | 0 | 0 | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0 | 6 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 6 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 1 | 1 | 6 | 4 | 2
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 4 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 5 | 5 | 3
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 3 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lividity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 4 | 0 | 0 | 2 | 1 | 3
Haematoma (Vascular disorders) | 3 | 0 | 0 | 1 | 2 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after first multi-site publication or if no multi-site publication is made within 18 months of study completion/termination. The only disclosure restriction on PI is sponsor can review results comms. prior to public release and can embargo comms. Regarding trial results for a period >60 but ≤180 days from time submitted to sponsor review. Sponsor can't require changes to the comms, extend embargo or require changes to comms, except removing confidential info that are not results.

DOCUMENTS (2):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT03684694/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT03684694/SAP_001.pdf